CLINICAL TRIAL: NCT03622398
Title: Highly Cross-linked Polyethylene Versus Compression Mold Conventional Polyethylene in Cruciate-substituting Total Knee Arthroplasty in Young Patients, a Randomized Trial
Brief Title: Highly Cross-linked Polyethylene in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Young Hoo Kim, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XPEPETKA
Record Dates: First submitted 2018-07-29; First posted 2018-08-09 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Knee Arthroplasty, Total
Keywords: total knee arthroplasty; highly cross-linked polyethylene
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Total knee arthroplasty is performed on patients with knee osteoarthritis. One group will receive a highly cross-linked polyethylene liner and one group will receive a conventional polyethylene liner. Other parts of procedures will be the same.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HXLPE (Experimental): This side of knee implanted with HXLPE(highly crosslinked polyethylene) liner while undergoing total knee arthroplasty. This group will receive the intervention, "Total knee arthroplasty with HXLPE liner".
  Interventions: Procedure: Total knee arthroplasty with HXLPE liner
- Conventional (Active Comparator): This side of knee implanted with conventional polyethylene while undergoing standard total knee arthroplasty. This group will receive the intervention, "Total knee arthroplasty with conventional polyethylene liner".
  Interventions: Procedure: Total knee arthroplasty with conventional polyethylene liner

INTERVENTIONS:
Procedure: Total knee arthroplasty with HXLPE liner — Replacing arthritic knee with a metal device, and using a highly cross-linked polyethylene(HXLPE) liner in between metallic surfaces.
  Arms: HXLPE
Procedure: Total knee arthroplasty with conventional polyethylene liner — Replacing arthritic knee with a metal device, and using a conventional polyethylene liner in between metallic surfaces.
  Arms: Conventional

SUMMARY:
The aim of this study was to determine clinical and radiographic results after posterior cruciate-substituting total knee arthroplasties with highly cross-linked polyethylene in one knee and compression mold conventional polyethylene in the contralateral knee in the same patients.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 65 years old
* with end stage knee arthritis bad enough for knee replacement

Exclusion Criteria:

* inflammatory arthritis
* combined foot and ankle disorders.
* dementia
* patient older than 65 years old.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Knee society knee score | minimum 10 year follow up after the index surgery
  a proven score for the measurement of knee function, the score ranges from 0 to 100, 100 being the best possible score, indicating normal knee function

SECONDARY OUTCOMES:
WOMAC(Western Ontario and McMaster Universities) Scores | minimum 10 year follow up after the index surgery
  A tool to evaluate patient function associated with knee. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). The total score is summed from individual sections, and 0 is the best possible score.
Range of motion | minimum 10 year follow up after the index surgery
  maximum flexion of the knee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim YH, Oh JH, Oh SH. Osteolysis around cementless porous-coated anatomic knee prostheses. J Bone Joint Surg Br. 1995 Mar;77(2):236-41. PMID 7706337
- [Background] Mikulak SA, Mahoney OM, dela Rosa MA, Schmalzried TP. Loosening and osteolysis with the press-fit condylar posterior-cruciate-substituting total knee replacement. J Bone Joint Surg Am. 2001 Mar;83(3):398-403. doi: 10.2106/00004623-200103000-00012. PMID 11263644
- [Background] Rodriguez JA, Bhende H, Ranawat CS. Total condylar knee replacement: a 20-year followup study. Clin Orthop Relat Res. 2001 Jul;(388):10-7. PMID 11451106
- [Background] Hodrick JT, Severson EP, McAlister DS, Dahl B, Hofmann AA. Highly crosslinked polyethylene is safe for use in total knee arthroplasty. Clin Orthop Relat Res. 2008 Nov;466(11):2806-12. doi: 10.1007/s11999-008-0472-4. Epub 2008 Sep 10. PMID 18781371
- [Background] Long WJ, Levi GS, Scuderi GR. Highly cross-linked polyethylene in posterior stabilized total knee arthroplasty: early results. Orthop Clin North Am. 2012 Nov;43(5):e35-8. doi: 10.1016/j.ocl.2012.07.005. Epub 2012 Sep 27. PMID 23102419